CLINICAL TRIAL: NCT00205946
Title: The Effects of Acute Administration of Bupropion on Neural Substrates Underlying Hedonic Capacity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affective Neuroscience Laboratory (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Diego Pizzagalli, Principal Investigator, Harvard University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-P-002234-1; 2004-P002234-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-11

CONDITIONS: Major Depressive Disorder
Keywords: Reward Processing; Wellbutrin; Bupropion
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bupropion (Active Comparator)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — 150 mg of bupropion administered 5 hours before fMRI scanning
  Other Names: Wellbutrin XL
  Arms: Bupropion
Drug: Placebo — Administered 5 hours prior to fMRI scanning (randomly assigned, double blind)
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effects of a single-dose of Wellbutrin XL (bupropion hydrochloride) on reward processing.

DETAILED DESCRIPTION:
A cardinal feature of Major Depressive Disorder is anhedonia, which is a lack of pleasure in normally enjoyable activities. In order to understand reward processing in depressed individuals it is also necessary to study reward processing in people who are not depressed. Bupropion, the active drug in the anti-depressant Wellbutrin XL, has been shown to increase brain reward functioning in animals. The goal of the present study is to investigate the effects of Wellbutrin XL administered to psychiatrically healthy individuals as they perform a computer task known to assess reward processing.

ELIGIBILITY:
Inclusion Criteria:

* Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse)
* Non-Smoker
* Right-handed (Chapman and Chapman 1987)
* Ability to provide informed consent

Exclusion Criteria:

* Predisposition to seizure (e.g. family history of a seizure disorder, history of head trauma) or current use of medications that lower the seizure threshold
* History or current diagnosis of anorexia or bulimia
* Alcohol or substance abuse within the past year
* Current usage of Wellbutrin or Zyban or other drugs that contain bupropion
* Recent discontinuation of alcohol or sedatives (including benzodiazepines)
* Use of (in the last 2 weeks) medications that may have antidepressant properties (ex. some herbal supplements)
* Known allergies to bupropion
* Currently lactating, pregnant or believe you are likely to be pregnant (enrolled subjects who are not using reliable contraception and have engaged in sexual intercourse since their last menstrual period will be given a self-administered pregnancy test.)
* Left-handed/ambidextrous
* Evidence of neurological illness
* Serious suicide or homicide risk

Concomitant medications other than those listed in the exclusion criteria will be considered on an individual basis. Oral contraceptives will be allowed.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Whether an acute dose of bupropion vs. placebo differentially affects the neurobiology and behavior of reward processing in depressed participants. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, PhD, Principal Investigator — Harvard University
Locations (2):
- United States (2):
  - The Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts
  - Affective Neuroscience Laboratory, Department of Psychology, Harvard University, Cambridge, Massachusetts